CLINICAL TRIAL: NCT02974348
Title: Assessment of Antimalaria Drugs Susceptibility Testing for an Effective Management of Infected Patients in Sub-Sahara Africa
Brief Title: Antimalaria Drugs Susceptibility Testing for an Effective Management of Infected Patients in Sub-Sahara Africa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Bamenda (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government); National Institute for Parasitic Disease, Chinese Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CASTEP
Record Dates: First submitted 2016-11-18; First posted 2016-11-28 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Drug Resistant Malaria Due to Plasmodium Falciparum
MeSH Terms: interventions — Acetaminophen; Amoxicillin; Quinine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- arm 1: Arthemeter-lumefantrine (Active Comparator): Arthemeter-lumefantrine (ART-LUM) is an antimalaria drug manufactured as fixed combination tablets, each containing 20 mg of artemether and 120 mg of lumefantrine. ART-LUM was administrated according to body weight as six consecutive doses: The first dose at diagnosis and the second dose eight hours later, 0- 24-48 hours
  Interventions: Drug: Arthemeter-lumefantrine
- arm 2 : Artesunate mefloquine (Active Comparator): Artesunate mefloquine (ASMQ) is an antimalaria drug administered as a combination of artesunate, 4 mg/kg/day, with mefloquine, 8 mg/kg/day orally once a day for 3 days or three times, at an interval of 24 hours (0 h - 24 h - 48 h).
  Interventions: Drug: Artesunate mefloquine
- arm 3 : Dihydroartemisinin piperaquine (Active Comparator): Dihydroartemisinin piperaquine (DHA-PQ ) is an antimalaria drug administered as a combination of dihydroartemisinin, 2.5 mg per kg, with piperaquine phosphate, 20mg per kg daily for 3 days or three times, at an interval of 24 hours
  Interventions: Drug: Dihydroartemisinin piperaquine
- Paracetamol (Other): Oral paracetamol is administered at of 50mg/kg body weight per day in three divided doses for fever exceeding 37.5oC.
  Interventions: Drug: Paracetamol
- Amoxicillin (Other): amoxicillin is an antibiotic administered at 50mg per kg body weight per day for seven days in the event of concomitant bacterial infection, absent on day 0 but present during the follow up.
  Interventions: Drug: Amoxicillin
- Quinine (Other): Quinine is an antimalarial recommended by the WHO and NMCP to be used as second line treatment for malaria. In this study, for cases of treatment failure with the artemisinin based combination therapies, quinine sulphate is administered as a second line or rescue drug at a dose of 25mg base per kg body weight per day in three divided doses for five days. The participant is then classified as ETF or LTF and excluded from the study.
  Interventions: Drug: Quinine

INTERVENTIONS:
Drug: Arthemeter-lumefantrine — Randomization codes were computer-generated by an offsite investigator and provided to a study nurse responsible for treatment allocation. All other study personnel were blinded to the treatment assignments, and patients were not informed of their treatment regimen. Participants from Group 1: AL, Group 2 : DHAP, Group3 : ASMQ were also given appointment card for days 1, 2, 3, 7, 14, 21, 28, 35 and 42 for clinical examination and blood smears. Blood was taken on filter paper on each of these visits.
  Other Names: Cofantrine®
  Arms: arm 1: Arthemeter-lumefantrine
Drug: Artesunate mefloquine — Artequin® is an antimalarial drug presented as infant co-formulation of two separate drugs
  Other Names: Artequin®
  Arms: arm 2 : Artesunate mefloquine
Drug: Dihydroartemisinin piperaquine — Malacur®. is an antimalarial drug presentad as co-formulation of two separate drugs
  Other Names: Malacur®
  Arms: arm 3 : Dihydroartemisinin piperaquine
Drug: Paracetamol — Paracetamol, is an antipyretic drug, presented as tablets or syrup in infants formulation
  Other Names: Paracetamol syrup
  Arms: Paracetamol
Drug: Amoxicillin — Amoxicillin is an antibiotic with no reported activity on plasmodium
  Other Names: Clamoxyl® 125 mg/5mL
  Arms: Amoxicillin
Drug: Quinine — quinine sulphate is an antimalaria drug administered as a second line or rescue drug
  Other Names: Quinine sulphate
  Arms: Quinine

SUMMARY:
The antimalarial drugs efficacy and safety study will be conducted in the Clinics and hospital of the Cameroon Development Corporation (CDC) Estates, Tiko Health District, located in a typical forest and rainfall area in the South West Region Cameroon. In this study, 350 children aged 6 months to 5 years who are found to have uncomplicated symptomatic malaria will be enrolled between October 2012 and March 2013. Participants will be randomized to receive one of the following medications.

(i) DHA+PQ : dihydroartemisinin, 2.5 mg per kg, plus piperaquine phosphate, 20mg per kg daily for 3 days; (ii) ART LUM : Artemether, 2mg per kg, plus lumefantrine 10mg, twice daily for 3 days; (iii) AS+MQ: artesunate, 4 mg/kg/day, with mefloquine, 8 mg/kg/day orally once a day for 3 days.

All study medications will be administered orally The Primary objective of this study are to compare the efficacy, safety and tolerability of orally administered artemether plus lumefantrine (ART+LUM), artesunate plus mefloquine (AS+MQ) and dihydroartemisinin plus piperaquine (DHA+PQ) combinations in the treatment of uncomplicated falciparum malaria in Cameroon in order to provide evidence that can be used to determining the optimum antimalaria treatment policy in Cameroon. The secondary objectives are as follows (i) To valuate the efficacy and safety of artemether plus lumefantrine (ART + LUM) and artesunate plus mefloquine (AS + MQ) versus dihydroartemisinin plus piperaquine (DHA + PQ) combination (ii) To compare the clearance of asexual parasites and gametocytes in each treatment arm (iii) To assess the clearance of fever (iv) Assess effect of each treatment arm on anemia This study is a randomized, double blinded clinical trial. After enrollment, participant will be randomized to one of the three treatment regimen. The treatment outcome will be assessed through a 42-day efficacy study. Participants who will exhibit early or late treatment failure and those with adequate clinical response and parasitological failure on day 14, 28 or 42 will be treated with quinine (25mg base per kg body weight per day in three divided doses for five days). In addition to antimalarial drugs oral paracetamol (50mg/kg body weight per day in three divided doses) will be administered for fever exceeding 37.5%. Polymerase Chain Reaction (PCR) -corrected 28 day and 42 day efficacy will be evaluated for each treatment episode.

DETAILED DESCRIPTION:
Malaria incidence has increased two- to three-folds over the past four decades, and nearly half the world's population now lives in regions endemic for malaria: In Asia, Africa, and South America. A global annual estimate of 300-500 clinical cases of malaria and mortality in the range of 1-2 million is reported, 90% of which occurs in sub-Saharan Africa. In Cameroon, malaria remains the number one public health problem with more than one million five hundred cases and three thousand one hundred and sixty two deaths in health facilities per year. Indeed, 45-50% of consultations, 23% of hospitalizations and 35% of deaths among children under 5 years are attributable to malaria Early diagnosis and treatment for malaria remain the most acceptable strategy for malaria control. Mortality is rising and approaching three million malarial deaths each year, in large parts because of increasing resistance to antimalarial drugs. The emergence and spread of P. falciparum resistance to conventional monotherapies such as chloroquine (CQ), amodiaquine (AQ), mefloquine (MQ), sulfadoxine-pyrimethamine (SP) resulted in the request of more effective and accessible antimalaria drugs to the entire population living in endemic areas.

In Cameroon, prior to 2002, CQ and SP were the first and second line antimalarial drugs respectively. Studies conducted in different ecological settings in Cameroon revealed marked decline of these drugs with 67% clinical failure for CQ alone . This led to an interim adoption of AQ by the Ministry of Public Health. A series of randomised, open controlled trial revealed that AQ was still effective when administered as monotherapy or in combination with SP since only 10.2 %, 13.6 % and 0% clinical failures were recorded for AQ, SP and SP+AQ respectively. However, studies conducted in Guinea Savannah showed decline rates of these antimalarials drugs with clinical failures of 40%, 20%, and 13.6% for AQ, SP and AQ+SP combination.

Widespread resistance of malaria parasite to these commonly available antimalaria drugs has necessitated country to review and deploy new antimalarial drug policies to ensure effective case management. The World Health Organization (WHO) currently recommends artemisinin-based combination therapies (ACTs) as the best first-line treatment for uncomplicated falciparum malaria, but studies to ensure that current regimens are optimal are incomplete. Artemisinine-based combination therapies (ACTs) are most preferred for their enhancement of efficacy and their potential to lower malaria incidence and the rate at which resistance emerges and spread\. Due to their rapid clearance time, treating early cases of uncomplicated malaria with ACTs may prevent its progression to severe malaria with consequent reduction in severe cases and malaria mortality rate. Although the National Malaria Control Programme (NMCP) of Cameroon adopted amodiaquine plus artesunate (AQ+AS) and arthemether plus lumefantrine (ART+LUM) for the treatment of uncomplicated malaria in 2004, there was no local data in support of the policy. In series of subtrials to constitute a database of anti-malarial drug efficacy in Cameroon, AQ was proposed to be the most rational partner of artesunate; likewise, a single arm study provided preliminary evidence of safety and efficacy of AQ+AS but with low statistical power to detect rare events and no PCR corrections to distinguish re-infection from recrudescence. Meta-analysis studies have shown ART-LUM to be highly effective and safe when the twice daily doses (total of six doses) are administered under supervision, but there are concerns that six doses of ART-LUM over three days may reduce compliance. Nevertheless, relatively few numbers of patients complained of physical fatigue during ART-LUM treatment but trials comparing it to order ACTs are few. AS+AQ combination is less expensive and subsidized by the Cameroonian Government, it is believed that its cure rate may be lower than that of ART-LUM because of parasite resistance to AQ and as such, its inclusion in ACTs is likely going to fail. In addition, the minor, transient side effects of AQ may lead to poor compliance and subsequent decline in AQ efficacy. In Southeast Asia, where P. falciparum is the most drug-resistant in the world, three-day artesunate-mefloquine treatment is generally the preferred treatment for uncomplicated malarial infection. Studies in Laos, suggest that artesunate plus mefloquine (AS-MQ) and ART-LUM combinations are both effective and are superior to CQ plus SP in the treatment of uncomplicated falciparum malaria. However, ASMQ has been limited by the high cost, the frequency of adverse effects associated with mefloquine, and the lack of a formulation combining both antimalarials in a single tablet. In addition, reduced efficacy of artesunate-mefloquine has been reported recently from the southeastern border of Thailand.

Artemether plus lumefantrine has fewer adverse effects but is also relatively expensive. A global analysis of a series of randomized studies of anti-malarial treatment efficacy conducted in Cameroon between 2003 and 2007 ART-LUM to be the most effective ACT with no treatment failure due to recrudescence (98.3% cure rate PCR corrected), followed by dihydroartemisinin-piperaquine with 92.7% cure rate. After PCR adjustment, 28 days cure rates was 91.7% for AS-SP 88.7% for artesunate-amodiaquine, and 76% for artesunate-chlorproguanil-dapsone. Clinical trials in Cambodia and Vietnam suggest that the dihydroartemisinin plus piperaquine (DHA+PQ) combination is highly effective against P. falciparum parasites with few adverse effect in both children and adult. In Cambodia, the 28-days cure rates were 98.6% in children and 92.3% in adult and in Vietnam, using dihydroartemisinin-piperaquine-trimethoprim combination, the 56-days cure rates in children and adults were 97-98% (Tran et al., 2004). In addition, it is relatively inexpensive compare to other ACTs, at 1 $ US per treatment course (Mutabingwa et al., 2005).

Therefore if it is demonstrated that DHA-PQ is an effective antimalaria in Cameroon, with fewer adverse effects in comparison to AS-MQ and ART-LUM, it may be an alternative treatment available to the Government of Cameroon with the advantages of being coformulated and available at lower cost than the other ACTs.

In order to determine the comparative efficacy and adverse effects profile of antimalaria in Cameroon, investigators propose to carry out an open randomised comparative clinical trial of the combination of oral arthemether plus lumefantrine (ART+LUM) and artesunate plus mefloquine (AS+MQ)versus dihydroartemisinine plus piperaquine (DHA+PQ) combinations in the treatment of uncomplicated malaria.

Primary objective :

The objective of this study is to compare the efficacy, safety and tolerability of orally administered arthemether plus lumefantrine (ART+LUM), artesunate plus mefloquine (AS+MQ) and dihydroartemisinin plus piperaquine (DHA+PQ) combinations in the treatment of uncomplicated falciparum malaria in Cameroon in order to provide evidence that can be used to determining the optimum antimalaria treatment policy in Cameroon.

Secondary objectives :

* To valuate the efficacy and safety of artemether plus lumefantrine (ART + LUM) and artesunate plus mefloquine (AS + MQ) versus dihydroartemisinin plus piperaquine (DHA + PQ) combination
* To compare the clearance of asexual parasites and gametocytes in each treatment group
* To assess the clearance of fever
* To assess effect of each treatment arm on anemia

STUDY SITE AND DESIGN It is a randomized clinical trial comparing the efficacy of oral dihydroartemisinin plus piperaquine to artemether plus lumefantrine and artesunate mefloquine combinations. The formulation of the test will be unilateral (Null hypothesis: DHA +PQ = ART+LUM or DHA + PQ = AS + MQ ; Alternative hypothesis: DHA +PQ > ART+LUM or DHA + PQ> AS + MQ) The trial will be conducted in a typical forest and rainfall area located in south-western Region of Cameroon. Patients will be recruited in the outpatient pediatric unit of satellite clinics and references hospital under Cameroon Development Corporation (CDC) administration, between October 2012 and March 2013

ELIGIBILITY

* Inclusion criteria : The inclusion criteria are; signs/symptoms of uncomplicated malaria including axillary temperature ≥ 37.5; monoinfection with Plasmodium falciparum; parasite count between 2000 and 200 000 per μl; haemoglobin level> 5 g/dL; absence of signs/symptoms of severe malaria or other diseases requiring drugs with antimalaria or antihistaminic activities; parent/guardian willingness to give their consent
* Exclusion criteria: Exclusion of patients with the following criteria; Chronic disease (HIV, malnutrition etc.), severe malaria, severe anaemia (haemoglobin level< 5 g/dL), respiratory distress, inability to drink, convulsion etc., history of allergie to test drugs; co-infection requiring drug with antihistaminic or antimalaria activities such as cotrimoxazole

SAMPLING AND SAMPLE SIZE:

The minimum participant per arm was calculated to be 50 in order to detect reduction of fever for at least 12 hrs, with the standard deviation of 18, and α and β values set at 0.05. However, the sample size will be increase by 10% in order to take account of individuals lost of follow-up. Therefore the total number of participants to be enrolled in this study is estimated to be at least 180 with 60 participants per treatment arm.

INITIAL EXAMINATION This will include a complete physical examination and blood sample analysis. After finger pricking, samples of capillary blood will be used to prepare two thick films, to determine haematocrit, to conduct the Rapid Diagnosis Testing (RDT), impregnate an isocode stix (50 µl for DNA extraction) by depositing a drop of blood on this filter paper while avoiding any contact with the finger. All slides, cassette and stix will be labelled with patient's individual code numbers and date of collection. They will be air dried and kept away from insects. The stix will be stored with a desiccant in individual plastic bag. The microscopy slides will be stained and kept in slides boxes. Parasite density will be counted on thick blood film stained with Giemsa then examined under the microscope. The reading will be on 200 leukocytes and the result will be expressed in number of asexual parasites per µl of blood by estimating the average white Blood Cell (WBC) count of 8000/µl of blood. Anemia will be assessed by the measurement of hematocrit in heparinized capillary tube, centrifuged for 5 minutes. Finger prick blood sample will be used to search for the Plasmodium falciparum Histidin Rich Protein 2 (HRP2).The mutations responsible for drug resistance will be identified on isolates of P. falciparum, collected on filter paper by molecular biology techniques

TREATMENT REGIMEN

Upon arrival to the health facility, patients who will meet the inclusion criteria and give their consent, will be randomly assigned to one of the following combination and doses: (i) DHA+PQ : dihydroartemisinin, 2.5 mg per kg, plus piperaquine phosphate, 20mg per kg daily for 3 days; (ii) ART+ LUM : Artemether, 2mg per kg, plus lumefantrine 10mg, twice daily for 3 days; (iii) AS+MQ: artesunate, 4 mg/kg/day, with mefloquine, 8 mg/kg/day orally once a day for 3 days.

All drugs will be administered with water except for ART-LUM, which will be given with milk to increase bioavailability. All doses will be administered under supervision. After drug ingestion, the patient will be observed for at least 30 minutes. Children who will vomit within this period will receive the same repeated doses. Patients with persistent vomiting will be withdrawn from the study. After the procedure patients will be given a schedule for routine follow-up visits. Parents/guardians will be informed to immediately return their children/ to the assessment team at any time during or outside the follow-up periods if symptoms return.

The personnel who will administer the doses will be different from those who will follow the patient up and examine the blood smears.

Rescue treatment:

Children who will exhibited early or late treatment failure and those with adequate clinical response and parasitological failure on day 14, 28. or 42 will be treated with quinine (25mg base per kg body weight per day in three divided doses for five days), in accordance with the Cameroon National Malaria Control Program and the WHO guidelines on antimalarial treatment. In addition to antimalarial drugs oral paracetamol (50mg/kg body weight per day in three divided doses) will be administered for fever exceeding 37.5oC. In the event of concomitant bacterial infection, absent on day 0 but present during the follow up, amoxicillin will be administered at 50mg per kg body weight per day for seven days

Non recommended treatment: antibiotics such as cotrimoxazole with antimalaria or antihistaminic activities.

MONITORING FOR SAFETY, PARASITOLOGICAL AND CLINICAL RESPONSES The clinical response will be monitored on days 1, 2, 3, 7, 14, 28 and D42. All patients will be followed up by means of home or facility visit. Therapeutic efficacy will be evaluated in relation to three major criteria: (1) the fever clearance time define as the time taken to attain a rectal temperature below 38°C (ii) The proportion of negative thick smears on days 7, 14, 28, D42 and (iii) the number of early (D1-D3) and late (D4-D42) treatment failures. The clinical and parasitological responses will be classified as early treatment failure, late treatment failure or adequate clinical and parasitological response according to the WHO definition. Other criteria include recrudescence of parasitemia, frequency of advert effects side (pruritus, fatigue, headache, dizziness, nausea, vomiting, diarrhea, skin rash, palpitation, bradycardia). Judging criteria will be evaluated by observers unaware of the treatment administered. Rectal temperature will be taken with an electronic thermometer. Side effects will be noted from the statements of parent/guardians. Parasite densities will be read against 1000 leukocytes.

FOLLOW-UP PROCEDURE

Follow-up schedule Patients will be assessed daily during the scheduled follow-up. Adverse effects will be assessed based on non-suggestive questioning by the investigators. After patient enrolment at D0, clinical assessment will be made on day 1, 2, 3, 7, 14, 28 and 42 as recommended in the WHO protocol. Patients will be advised to return on any day outside the schedule period (D8-D13) (D15-D27), and (D29-D41) if symptoms returned and not to wait for scheduled visits. Blood films for parasite count and filters paper samples will be examined on these days or on any other day when ever a child spontaneously returns. Routine blood investigations (hematology and biochemistry) will be performed prior to (Day0) and weekly for the 4 weeks of the study period. Haemoglobin will be typically reassessed on day 7, 14, 28, 42. Provision will be made ahead of time for locating patients at home if they do not respond to schedules Study end-point Valid end point includes treatment failure, completion of follow-up period without treatment failure, loss of follow-up, protocol violation and severe adverse effects.

Statistical analysis The data will be analysed by means of Statistical Package for the Social Sciences (SPSS). Qualitative variables will be compared using the X2 or Fisher's exact test, and quantitative variables will be compared by analysis of variance or the Kruskaul-Wallis test. The 95% confidence intervals of proportions will be calculated using the binomial test and the level of significance (P) set at 0.05 for all statistical tests.

ETHICAL CONSIDERATION Tests drugs are included in national guidelines and are prescribed daily in Cameroon. The aim of the study, the advantages and the constraints will be explained in order to obtain the parent/guardian consent. Participation fee for all patients (transportation, laboratory analysis) will be free of charge.

Data collection and analysis

Data will be collected on separate standardized questionnaires for enrollment and monitoring. Follow-up questionnaires and patient case record forms will be handed to the coordinator on daily basis, who will archive them after verification and data analysis.

Estimated Time to Complete Enrollment:

The total duration of the survey is estimated at 150 days based on 83 days of enrolment (an average of 4 enrolments per day), 42 days for the follow-up of the last enrolled patient, and 25 days for data analysis and report writing.

ELIGIBILITY:
Inclusion Criteria:

* signs/symptoms of uncomplicated malaria with axillary temperature ≥ 37.5;
* monoinfection with Plasmodium falciparum;
* parasite count between 2000 and 200 000 per μl;
* haemoglobin level> 5 g/dL;
* absence of signs/symptoms of severe malaria or other diseases requiring drugs with antimalaria or antihistaminic activities;
* parent/guardian willingness to give their consent

Exclusion Criteria:

* Chronic disease (HIV, malnutrition etc.),
* severe anaemia (haemoglobin level< 5 g/dL),
* respiratory distress, inability to drink, convulsion etc.,
* history of intolerance to test drugs;
* co-infection requiring drug with antihistaminic or antimalaria activities such as cotrimozaxole

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
efficacy and safety assessment | 42 days
  The primary endpoint was the 28-day and 42-day cure rates and was defined as proportion of patients with adequate clinical and parasitological response (ACPR) after 28 and 42 days of follow-up. Absence of parasitemia until day 28 and day 42 irrespective of axillary temperature was categorized as an adequate clinical and parasitologic response (ACPR). Secondary endpoints were early treatment failure (ETF), late clinical failure (LCF), late parasitological failure (LPF), adverse events (clinical and laboratory abnormalities), anaemia (Hematocrit < 30%), clearance rate of fever and parasitaemia, and gametocyte

SECONDARY OUTCOMES:
Hemoglobin level | 42 days follow-up
  The ability of the drug to restore hemoglobin level back to normal
parasite clearance rate assessment | 42 days
  The ability of the drug to completely eliminate plasmodium in the blood stream including participant without symptoms of fever
PCR-correction | 42 days
  blood sample from patients with parasitaemia at any day of follow-up are analysed by PCR to evaluated the genetic profile of the MSP1 and MSP2

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonong Zhou, PhD, Study Director — National Institute for Parasitic Disease
Locations (1):
- CDC Hospital, Tiko, South-West Region, Cameroon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashley EA, White NJ. Artemisinin-based combinations. Curr Opin Infect Dis. 2005 Dec;18(6):531-6. doi: 10.1097/01.qco.0000186848.46417.6c. PMID 16258328
- [Background] Basco LK, Same-Ekobo A, Ngane VF, Ndounga M, Metoh T, Ringwald P, Soula G. Therapeutic efficacy of sulfadoxine-pyrimethamine, amodiaquine and the sulfadoxine-pyrimethamine-amodiaquine combination against uncomplicated Plasmodium falciparum malaria in young children in Cameroon. Bull World Health Organ. 2002;80(7):538-45. PMID 12163917
- [Background] Brasseur P, Druilhe P, Kouamouo J, Brandicourt O, Danis M, Moyou SR. High level of sensitivity to chloroquine of 72 Plasmodium falciparum isolates from southern Cameroon in January 1985. Am J Trop Med Hyg. 1986 Jul;35(4):711-6. doi: 10.4269/ajtmh.1986.35.711. PMID 3524286
- [Background] Tran TH, Dolecek C, Pham PM, Nguyen TD, Nguyen TT, Le HT, Dong TH, Tran TT, Stepniewska K, White NJ, Farrar J. Dihydroartemisinin-piperaquine against multidrug-resistant Plasmodium falciparum malaria in Vietnam: randomised clinical trial. Lancet. 2004 Jan 3;363(9402):18-22. doi: 10.1016/s0140-6736(03)15163-x. PMID 14723988
- [Background] Breman JG, Alilio MS, Mills A. Conquering the intolerable burden of malaria: what's new, what's needed: a summary. Am J Trop Med Hyg. 2004 Aug;71(2 Suppl):1-15. PMID 15331814
- [Background] Djimde A, Doumbo OK, Cortese JF, Kayentao K, Doumbo S, Diourte Y, Coulibaly D, Dicko A, Su XZ, Nomura T, Fidock DA, Wellems TE, Plowe CV. A molecular marker for chloroquine-resistant falciparum malaria. N Engl J Med. 2001 Jan 25;344(4):257-63. doi: 10.1056/NEJM200101253440403. PMID 11172152
- [Background] Mangham LJ, Cundill B, Achonduh OA, Ambebila JN, Lele AK, Metoh TN, Ndive SN, Ndong IC, Nguela RL, Nji AM, Orang-Ojong B, Wiseman V, Pamen-Ngako J, Mbacham WF. Malaria prevalence and treatment of febrile patients at health facilities and medicine retailers in Cameroon. Trop Med Int Health. 2012 Mar;17(3):330-42. doi: 10.1111/j.1365-3156.2011.02918.x. Epub 2011 Nov 21. PMID 22098135
- [Background] Mbacham W.F., Njuabe MT., Evehe MS., Moyou R., Skobo A., (2005a) Antimalarial drug studies in Cameroon reveal deteriorating fansidar and amodiaquine cure rates. Malaria research and control in Cameroon.. J. Cam. Acad. Sci., 5 : 58-63.
- [Background] Mbacham W, Evehe M, Mbulli A, Akaragwe I, Tawe B, Djoko C, Gang B, Masumbe P, Mokube A, Atogho B, Ebeng R. (2005b) Therapeutic efficacy of Sulfadoxine-Pyrimethamine (Fansidar®) and mutation rates to Anti-folate genes in different regions of Cameroon. Acta Trop, 95S:337.
- [Background] Murray CJ, Rosenfeld LC, Lim SS, Andrews KG, Foreman KJ, Haring D, Fullman N, Naghavi M, Lozano R, Lopez AD. Global malaria mortality between 1980 and 2010: a systematic analysis. Lancet. 2012 Feb 4;379(9814):413-31. doi: 10.1016/S0140-6736(12)60034-8. PMID 22305225
- [Background] Mutabingwa TK. Artemisinin-based combination therapies (ACTs): best hope for malaria treatment but inaccessible to the needy! Acta Trop. 2005 Sep;95(3):305-15. doi: 10.1016/j.actatropica.2005.06.009. PMID 16098946
- [Background] NMCP (2007). National Malaria Control Program malaria report 2007.
- [Background] Ringwald P, Keundjian A, Same Ekobo A, Basco LK. [Chemoresistance of Plasmodium falciparum in the urban region of Yaounde, Cameroon. Part 2: Evaluation of the efficacy of amodiaquine and sulfadoxine-pyrimethamine combination in the treatment of uncomplicated Plasmodium falciparum malaria in Yaounde, Cameroon]. Trop Med Int Health. 2000 Sep;5(9):620-7. doi: 10.1046/j.1365-3156.2000.00614.x. French. PMID 11044276
- [Background] Snow RW, Guerra CA, Noor AM, Myint HY, Hay SI. The global distribution of clinical episodes of Plasmodium falciparum malaria. Nature. 2005 Mar 10;434(7030):214-7. doi: 10.1038/nature03342. PMID 15759000
- [Background] Soula G. , Ndounga M., Foumane V., Olivier G., Youmba J.C. Basco L. K., Boudin C., Same Ekobo A.., Ringwald P. (2000). Bilan de la résistance de P. falciparum à la chloroquine au Cameroun et alternatives thérapeutiques. Bull.liais. doc. OCEAC : 33(4) : 13-22.
- [Background] Silachamroon U, Krudsood S, Thanachartwet W, Tangpukdee N, Leowattana W, Chalermrut K, Srivilairit S, Wilaiaratana P, Thimasarn K, Looareesuwan S. An open, randomized trial of three-day treatment with artesunate combined with a standard dose of mefloquine divided over either two or three days, for acute, uncomplicated falciparum malaria. Southeast Asian J Trop Med Public Health. 2005 May;36(3):591-6. PMID 16124422
- [Background] Smithuis F, Kyaw MK, Phe O, Aye KZ, Htet L, Barends M, Lindegardh N, Singtoroj T, Ashley E, Lwin S, Stepniewska K, White NJ. Efficacy and effectiveness of dihydroartemisinin-piperaquine versus artesunate-mefloquine in falciparum malaria: an open-label randomised comparison. Lancet. 2006 Jun 24;367(9528):2075-85. doi: 10.1016/S0140-6736(06)68931-9. PMID 16798391
- [Background] Staedke SG, Kamya MR, Dorsey G, Gasasira A, Ndeezi G, Charlebois ED, Rosenthal PJ. Amodiaquine, sulfadoxine/pyrimethamine, and combination therapy for treatment of uncomplicated falciparum malaria in Kampala, Uganda: a randomised trial. Lancet. 2001 Aug 4;358(9279):368-74. doi: 10.1016/S0140-6736(01)05557-X. PMID 11502317
- [Background] Vijaykadga S, Rojanawatsirivej C, Cholpol S, Phoungmanee D, Nakavej A, Wongsrichanalai C. In vivo sensitivity monitoring of mefloquine monotherapy and artesunate-mefloquine combinations for the treatment of uncomplicated falciparum malaria in Thailand in 2003. Trop Med Int Health. 2006 Feb;11(2):211-9. doi: 10.1111/j.1365-3156.2005.01557.x. PMID 16451346
- [Background] Whegang SY, Tahar R, Foumane VN, Soula G, Gwet H, Thalabard JC, Basco LK. Efficacy of non-artemisinin- and artemisinin-based combination therapies for uncomplicated falciparum malaria in Cameroon. Malar J. 2010 Feb 19;9:56. doi: 10.1186/1475-2875-9-56. PMID 20170477
- [Background] World Health Organization. Guidelines for the treatment of malaria. 1st ed. Geneva: WHO, 2006.
- [Background] World malaria Report (2011). Global malaria incidence and Mortality rates
- [Background] Zikusooka CM, McIntyre D, Barnes KI. Should countries implementing an artemisinin-based combination malaria treatment policy also introduce rapid diagnostic tests? Malar J. 2008 Sep 15;7:176. doi: 10.1186/1475-2875-7-176. PMID 18793410
- [Derived] Metoh TN, Chen JH, Fon-Gah P, Zhou X, Moyou-Somo R, Zhou XN. Genetic diversity of Plasmodium falciparum and genetic profile in children affected by uncomplicated malaria in Cameroon. Malar J. 2020 Mar 18;19(1):115. doi: 10.1186/s12936-020-03161-4. PMID 32188442